CLINICAL TRIAL: NCT03526497
Title: Correlation Between Peripheral Venous Pressure and Central Venous Pressure in the Cardiac Intensive Care Unit
Status: Terminated | Type: Observational
Why Stopped: Poor enrollment
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 18-325
Record Dates: First submitted 2018-04-05; First posted 2018-05-16 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Prospective Studies; Heart Failure
Keywords: Catheterization, Peripheral/methods; Humans; Acute Disease; Aged; Female; Male; Follow-Up Studies; Heart Failure/physiopathology; Prospective Studies; Stroke Volume/physiology; Venous Pressure/physiology
MeSH Terms: conditions — Heart Failure; Acute Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In patients admitted to a coronary care unit, what is the correlation coefficient and limits of agreement for paired measurements of peripheral venous pressure and central venous pressure at multiple time points during the patient's hospitalization?

DETAILED DESCRIPTION:
The treatment of numerous cardiac conditions requires assessment of intravascular volume status, using central venous pressure (CVP) as the gold standard. Measurement of CVP requires placement of an invasive venous catheter, with insertion of a venous catheter into a central vein to obtain CVP. Catheter placement is invasive, costly and not without complications. Ideally, there would exist a peripheral surrogate for CVP that would be 1) minimally invasive to obtain, 2) low cost and 3) strongly correlate with CVP over a wide range of physiological conditions.

The peripheral venous system is in continuity with the central venous system and, as such, would be expected to have a pressure that correlates with central venous pressure. Numerous previous studies suggest a correlation between peripheral venous pressure (PVP) and central venous pressure. Prior studies have demonstrated a reasonable correlation between CVP and PVP in patient populations including decompensated heart failure, cardiac and non-cardiac surgery(1), liver transplant donors(2) and recipients(3), neurosurgical(4) and pediatric patients.(5) In an earlier study published by the authors of this paper, the mean difference between PVP and CVP in patients with acute heart failure syndromes was 0.4 mmHg with a correlation coefficient of 0.947. One limitation of the earlier study was that it established this correlation at only one point in time. In the study presented here, PVP and CVP will be obtained and correlation will be assessed across multiple time points during a given patient's hospitalization.

This is a prospective, single center cohort study to investigate the correlation between peripheral venous pressure and central venous pressure.

ELIGIBILITY:
Inclusion Criteria:

* We plan to enroll patients who meet the following criteria: Patients admitted to an intensive care unit for invasive hemodynamic monitoring. All eligible patients will be those who have already undergone pulmonary artery catheterization via the internal jugular or subclavian veins and upper extremity peripheral IV placement per routine standard of care prior to enrollment.

Exclusion Criteria:

* Patients will be excluded from this study for the following reasons: age less than 18 years of age, inability to obtain consent, femoral pulmonary artery catheter, or if their attending physician refuses to allow enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with pulmonary artery catheters and peripheral IVs admitted to the Coronary Care Units at the Cleveland Clinic, meeting the inclusion criteria, will be considered for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
In patients admitted to a coronary care unit, what is the correlation coefficient and limits of agreement for paired measurements of PVP and CVP at multiple time points during the patient's hospitalization? | 7-14 days
  Peripheral Venous Pressure and Central Venous pressure will be measured at three time points across a patient's hospitalization. The correlation coefficient and limits of agreement for paired measurements will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Mazen Hanna, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States